CLINICAL TRIAL: NCT01840475
Title: International, Multicenter, Non-interventional, Prospective, Longitudinal Study to Investigate the Effectiveness of Botulinum Toxin A (Dysport®) Injections in Patients Suffering From Post-stroke Arm Spasticity With Respect to Early, Medium or Late Start of Treatment.
Brief Title: Arm Spasticity - Non-Interventional Study Early BIRD (BoNT Treatment: Initial and Repeated Documentation)
Acronym: EARLYBIRD
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-94-52120-174
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Post-stroke Arm Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Botulinum toxin type A (BoNT-A) injection (Dysport®) Naïve: Subjects naïve to BoNT-A treatment.
- Botulinum toxin type A (BoNT-A) Pre-treated: Subjects pre-treated with BoNT-A.
  Investigators follow their individual injection protocol for the treatment with BoNT-A (modalities of administration in accordance with local Summary of Product Characteristics [SmPC]).

SUMMARY:
Botulinum toxin A (BoNT-A) is effective and safe in alleviating post-stroke spasticity and reducing the burden of associated symptoms.

The hypothesis for this non-interventional study in arm spasticity (AS-NIS early BIRD) is no significant difference between naïve and pre-treated patients. The patients will be divided in sub-groups according to the time interval between occurrence of stroke and start of treatment (early, medium and late start of treatment according to the first and third quartiles time distribution). It is hypothesized that the "early" start of treatment group will have a reduced modified Ashworth scale (MAS) on the elbow and wrist flexors when compared to the "late" start of treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to data collection
* Hemiparesis and clinically relevant upper limb post-stroke spasticity
* Treated with Dysport® or with the intention to be treated with Dysport® according to local SmPC
* BoNT naïve or pre-treated with any BoNT product

Exclusion Criteria:

* Recurrent stroke
* Sensitivity to Dysport® or to its excipients or any other contraindications as given in the local SmPC for Dysport®

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from post-stroke arm spasticity registered with Neurological clinics, Rehab centers with BoNT out-patient clinics and neurological practices.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2013-03; Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
Comparison of modified Ashworth scale (MAS) between patients with early start of treatment and patients with late start of treatment in the overall population (naive and pre-treated). | Final study visit: approximately 20 months after first visit
  "Early" and "late" start of treatment according to the first and third quartiles time distribution between stroke and start of treatment with BoNT-A.
  Investigation of effectiveness of BoNT-A treatment on the evolution of spasticity using MAS (sum of elbow and wrist flexors, EWF).

SECONDARY OUTCOMES:
Comparison of modified Ashworth scale (MAS) between patients with early start of treatment and patients with late start of treatment in the overall population (naive and pre-treated). | Approximately every 4 months starting from baseline up to 2 years
  "Early" and "late" start of treatment according to the first and third quartiles time distribution between stroke and start of treatment with BoNT-A.
  Investigation of effectiveness of BoNT-A treatment on the evolution of spasticity using MAS (sum of elbow and wrist flexors, EWF).

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (5):
- Hermagor, Austria
- Bidart, France
- Berlin, Germany
- Zwolle, Netherlands
- Bern, Switzerland